CLINICAL TRIAL: NCT00537082
Title: A 6-month, Double-blind, Randomized, Placebo-controlled, Parallel-group, Multicenter Study Comparing Efficacy and Safety of FTY720 0.5 mg and 1.25 mg Administered Orally Once Daily in Patients With Relapsing Multiple Sclerosis
Brief Title: Efficacy and Safety of FTY720 in Patients With Relapsing Multiple Sclerosis (MS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Collaborators: Tanabe Pharma Corporation (Industry)
Responsible Party: External Affairs
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CFTY720D1201
Record Dates: First submitted 2007-09-26; First posted 2007-09-28 (Estimated); Results first posted 2011-03-23 (Estimated); Last update posted 2011-04-21 (Estimated); Status verified 2011-04

CONDITIONS: Multiple Sclerosis
Keywords: FTY720,; MS
MeSH Terms: conditions — Multiple Sclerosis | interventions — Fingolimod Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (3):
- FTY720 0.5 mg (Experimental): FTY720
  Interventions: Drug: FTY720
- FTY720 1.25 mg (Experimental): FTY720
  Interventions: Drug: FTY720
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: FTY720 — Administered orally once daily for 6 months
  Arms: FTY720 0.5 mg; FTY720 1.25 mg
Drug: Placebo — Administered orally once daily for 6 months
  Arms: Placebo

SUMMARY:
To provide efficacy and safety data of two doses (0.5 mg and 1.25 mg) of FTY720 in Japanese patients with relapsing multiple sclerosis (MS)

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 18-60
* Patients with a diagnosis of multiple sclerosis

Exclusion Criteria:

* Patients with a history or presence of chronic disease of the immune system other than MS
* Patients with a history or presence of malignancy, pulmonary or heart disease, etc.
* Pregnant or nursing (lactating) women

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 171 (Actual)
Dates: Start 2007-09; Primary Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Japan, Principal Investigator — +81 3 3797 8748
Locations (15):
- Japan (15):
  - Novartis Investigative site, Sapporo, Hokkaido
  - Novartis Investigative Site, Chiba
  - Novartis Investigative Site, Ehime
  - Novartis Investigative Site, Fukuoka
  - Novartis Investigative Site, Gunma
  - Novartis Investigative Site, Hyōgo
  - Novartis Investigative Site, Ibaraki
  - Novartis Investigative Site, Kanagawa
  - Novartis Investigative Site, Kyoto
  - Novartis Investigative Site, Niigata
  - Novartis, Numakunai
  - Novartis Investigative Site, Osaka
  - Novartis Investigative Site, Tochigi
  - Novartis Investigative Site, Tokyo
  - Novartis Investigative Site, Wakayama

REFERENCES:
- [Derived] Saida T, Itoyama Y, Kikuchi S, Hao Q, Kurosawa T, Ueda K, Auberson LZ, Tsumiyama I, Nagato K, Kira JI. Long-term efficacy and safety of fingolimod in Japanese patients with relapsing multiple sclerosis: 3-year results of the phase 2 extension study. BMC Neurol. 2017 Jan 28;17(1):17. doi: 10.1186/s12883-017-0794-5. PMID 28129749
- [Derived] Saida T, Kikuchi S, Itoyama Y, Hao Q, Kurosawa T, Nagato K, Tang D, Zhang-Auberson L, Kira J. A randomized, controlled trial of fingolimod (FTY720) in Japanese patients with multiple sclerosis. Mult Scler. 2012 Sep;18(9):1269-77. doi: 10.1177/1352458511435984. Epub 2012 Feb 21. PMID 22354739

RESULTS

PARTICIPANT FLOW:
Groups:
- FTY720 1.25 mg; FTY720 0.5 mg; Placebo: Administered orally once daily for 6 months
Period: Overall Study
Arm/Group | FTY720 1.25 mg | FTY720 0.5 mg | Placebo
Started | 57 | 57 | 57
Completed | 48 | 48 | 51
Not Completed | 9 | 9 | 6
Not completed — Adverse Event | 6 | 6 | 3
Not completed — Protocol Violation | 0 | 2 | 1
Not completed — Lack of Efficacy | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Discontinued before initiating treatment | 3 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FTY720 1.25 mg | FTY720 0.5 mg | Placebo | Total
Number analyzed (Participants) | 57 | 57 | 57 | 171
Age Continuous [Mean (Standard Deviation); unit: years] | 36.0 (9.31) | 35.0 (9.01) | 35.0 (8.93) | 35.3 (9.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 40 | 39 | 118
  Male | 18 | 17 | 18 | 53
Region of Enrollment [Number; unit: participants]
  Japan | 57 | 57 | 57 | 171

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Free of Gadolinium-enhanced T1-Weighted Magnetic Resonance Imaging (MRI) Lesions at Both Month 3 and Month 6
Description: Brain Magnetic Resonance Imaging (MRI) was performed at Month 3 and Month 6. Gadolinium-enhancing lesions (active lesions) represent acute inflammatory activity only and dissipate within 2-8 weeks of appearance. MRI scans were analyzed by blinded readers at the central MRI Evaluation Center to ensure consistency. Any Gd-enhanced T1 weighted MRI data obtained less than 14 days after the steroid used to treat MS relapses is invalid and excluded.
Time Frame: Month 3 and Month 6
Population: Modified Full Analysis Set (Modified FAS) included all patients who were randomized and received at least one dose of study drug and had at least one valid post-randomized MRI scan at Month 3 or longer.
Measure: Number; unit: Participants
Arm/Group | FTY720 1.25 mg | FTY720 0.5 mg | Placebo
Number analyzed (Participants) | 50 | 50 | 52
Participants | 43 | 35 | 21

2. Secondary Outcome: Number of Patients Free of MS Relapse up to Month 6 (Confirmed Relapse Only)
Description: A relapse must have been confirmed by a neurologist and was confirmed when it was accompanied by an increase of at least half a step (0.5) on the Expanded Disability Status Scale (EDSS) or an increase of 1 point on two different Functional Systems (FS) of the EDSS or 2 points on one of the FS (excluding Bowel/Bladder or Cerebral FS).
Time Frame: up to Month 6
Population: Full Analysis Set (FAS) consisted of all patients who were randomized and received at least one dose of study drug. This population was only used for the analyses of relapse and EDSS.
Measure: Number; unit: Participants
Arm/Group | FTY720 1.25 mg | FTY720 0.5 mg | Placebo
Number analyzed (Participants) | 54 | 57 | 57
Participants | 45 | 45 | 37

3. Secondary Outcome: Number of Patients Free of New or Newly Enlarged T2 Lesions
Description: The number of T2 lesions were obtained from MRI scans at Screening visit. The numbers of new/newly enlarging T2 lesions were obtained from MRI scans at Month 3 or more. New lesions were identified by comparing each lesion already seen in previous examinations. Lesions expanding throughout several slices were counted as only one lesion.
Time Frame: up to Month 3 and up to Month 6
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | FTY720 1.25 mg | FTY720 0.5 mg | Placebo
Number analyzed (Participants) | 50 | 50 | 52
Participants
  Month 3 (n = 50, 49, 51) | 30 | 34 | 23
  Month 6 (n = 48, 48, 50) | 28 | 31 | 18

4. Secondary Outcome: Annualized Relapse Rate (ARR) at 6 Months
Description: Annualized relapse rate (ARR) of the treatment group is calculated by taking the total number of confirmed relapses for all the patients in the treatment group divided by the total number of days on study for all patients in the group and multiplied by 365.25 to obtain the annual rate.
Time Frame: 6 Months
Population: as for outcome 2
Measure: Number; unit: Relapses per year
Arm/Group | FTY720 1.25 mg | FTY720 0.5 mg | Placebo
Number analyzed (Participants) | 54 | 57 | 57
Relapses per year | 0.407 | 0.512 | 1.131

ADVERSE EVENTS:
Groups:
- FTY720 1.25mg; FTY720 0.5mg; Placebo: Administered orally once daily for 6 months
Arm/Group | FTY720 1.25mg | FTY720 0.5mg | Placebo
Serious Adverse Events (participants affected / at risk) | 11/54 | 5/57 | 3/57
Other Adverse Events (participants affected / at risk) | 42/54 | 41/57 | 27/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FTY720 1.25mg (N=54) | FTY720 0.5mg (N=57) | Placebo (N=57)
Atrioventricular block first degree (Cardiac disorders) | 0 | 1 | 0
Atrioventricular block second degree (Cardiac disorders) | 2 | 0 | 0
Bradycardia (Cardiac disorders) | 8 | 3 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0
Stress cardiomyopathy (Cardiac disorders) | 0 | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 1
Chest discomfort (General disorders) | 0 | 1 | 0
Malaise (General disorders) | 0 | 1 | 0
Heart rate decreased (Investigations) | 1 | 0 | 0
Liver function test abnormal (Investigations) | 1 | 0 | 0
Facial palsy (Nervous system disorders) | 1 | 0 | 0
Multiple sclerosis relapse (Nervous system disorders) | 1 | 0 | 0
Abortion induced (Surgical and medical procedures) | 0 | 0 | 1
Hypotension (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | FTY720 1.25mg (N=54) | FTY720 0.5mg (N=57) | Placebo (N=57)
Leukopenia (Blood and lymphatic system disorders) | 3 | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 3 | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 4 | 1
Dental caries (Gastrointestinal disorders) | 3 | 3 | 1
Diarrhoea (Gastrointestinal disorders) | 6 | 3 | 3
Gastritis (Gastrointestinal disorders) | 3 | 2 | 0
Nausea (Gastrointestinal disorders) | 5 | 4 | 2
Pyrexia (General disorders) | 2 | 2 | 4
Bronchitis (Infections and infestations) | 3 | 1 | 0
Nasopharyngitis (Infections and infestations) | 21 | 24 | 19
Pharyngitis (Infections and infestations) | 3 | 3 | 3
Tinea pedis (Infections and infestations) | 1 | 3 | 2
Liver function test abnormal (Investigations) | 18 | 12 | 3
Dizziness (Nervous system disorders) | 3 | 4 | 1
Headache (Nervous system disorders) | 5 | 5 | 4
Rash (Skin and subcutaneous tissue disorders) | 2 | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.